CLINICAL TRIAL: NCT04034030
Title: Repeated Oscillatory Transcranial Magnetic Stimulation Therapy of the Epileptogenic Cortical Area in Children With Focal Continuous-Spike and Wave During Sleep
Brief Title: Repeated Oscillatory TMS Therapy of the Epileptogenic Cortical Area in Children With Focal CSWS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Cornell University (Other)
Responsible Party: Principal Investigator, Lalit Bansal, Principal Investigator, Children's Mercy Hospital Kansas City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000245
Record Dates: First submitted 2019-07-22; First posted 2019-07-26 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: CSWS
Keywords: magnetic brain stimulation
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment Group (Experimental): This study will be conducted over one year in 10 focal CSWS patients ranging in age from 3 to 21 years. The patients will be recruited from the large patient population that is served by the Children's Mercy Comprehensive Epilepsy Monitoring Unit (EMU) in Overland Park, Kansas. Subjects will be identified from these EMU patient population. Those meeting inclusion criteria will be approached for possible enrollment. Inclusion criteria will be defined by patients that were diagnosed with focal CSWS in accordance with the ILAE classification with SWI >85% during NREM sleep on their previous or most recent EEG. Patients and their parents/guardians will provide assent/consent for participation in the study after being briefed on the nature of the study, by reading and signing assent and assent/consent forms, respectively
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Each patient will receive a 10 minute treatment of one time stimulation of the Epileptogenic Cortical Area (ECA). The TRPMS cap will be worn over the previously fixed scalp EEG electrodes. The procedure during this treatment session will consist of positioning a device microstimulator component centered on an area of focal epileptiform discharges (identified with EEG electrode placement) with the patient relaxing in a chair.
  The stimulus parameters used will be 120 stimulus trains of 100 ms in duration, each train delivered every 5 s for total session duration of 10 min. . The investigators will measure the subject for adequate placement of the device prior to stimulation. Once the placement of the device is confirmed, the study technician administrating the treatment will turn on the device using the app downloaded on an electronic device connected by Bluetooth to the device.
  Other Names: Trancranial Rotating Permanent Magnet Stimulator (TRPMS)

SUMMARY:
The investigators are investigating the effectiveness of a wearable multisite transcranial magnetic stimulation (mTMS) device that can deliver stimuli at multiple cortical sites simultaneously or sequentially for the treatment of an epileptic syndrome - focal continuous-spike and wave during sleep.

DETAILED DESCRIPTION:
Continuous Spike and Wave during Sleep (CSWS) is a rare neurological disease with an incidence of 0.2 - 0.5% of childhood epilepsy. It is often accompanied by comprehensive damage to brain function and associated neurodevelopmental problems. It is an epileptic syndrome which seriously affects the cognitive function of children. While it can be treated with drugs, other modalities are being sought, especially, in cases that are resistant to standard treatment. One such approach that is being tested is repetitive magnetic stimulation (rTMS). Noninvasive magnet stimulation of the cerebral cortex is an important and useful technique in neuroscience research, as well as in diagnostic and therapeutic clinical investigations. Over the last three decades the magnetic stimulation procedure is being carried out using a device called transcranial magnetic stimulator (TMS), which uses a large hand-held electromagnetic coil passing high amplitude current to induce her rapid changing magnetic field at a single cortical site. TMS has found clinical application several neurological and psychiatric conditions such as stroke, major depression, migraine, movement disorders and Tourette syndrome. One limitation of conventional TMS, besides the bulkiness of the device and large amount of current involved, is that it allows stimulation at only one cortical site at a time.Dr. Santosh Helekar of Houston Methodist Research Institute (HMRI) and Dr. Henning Voss of Weill-Cornell Medical College (WCMC) have developed a compact portable and wearable multisite transcranial magnetic stimulation device called Transcranial Rotating Permanent Magnet Stimulator (TRPMS) that can deliver stimuli at multiple cortical sites simultaneously or sequentially. It uses rapidly rotating small high-strength permanent magnets to induce currents in the brain. As opposed to conventional TMS, the TRPMS device is also ideally suited to conduct double blinded placebo controlled studies because undetectable demagnetized magnets can be intermixed with actual magnet to allow rapid rotation of either type of magnets to be activated and one in the same device in a randomized protocol. Under a previously approved HMRI study protocol this new device has been shown to induce motor-evoked potentials (MEPs) in the thenar muscles by highly focused stimulation of the cortical representation in the precentral gyrus.

In the present study, the investigators would like to conduct a test to see the therapeutic effectiveness of focused TRPMS stimulation of the epileptogenic region found on scalp electroencephalogram (EEG) in patients with focal CSWS. The specific aim of the study are:

1. To look at the immediate benefit obtained by CSWS patients subjected to 10 minutes of one-time TRPMS-ECA (epileptogenic cortical area) stimulation; evaluated as a reduction in Spike-Wave Index (SWI) on EEG during sleep.
2. To look at duration of sustainability (hours) of change in SWI achieved post stimulation.
3. To look at the tolerability of patients in using TRPMS.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 3 and 21 years old,
* An electroclinical diagnosis of focal CSWS as defined by ILAE
* SWI of ≥ 85% in sleep on EEG's performed on previous or most recent EEG study.
* No change in antiepileptic drugs (AED) in last 2 week, or patients not on any AED

Exclusion Criteria:

* Presence of metal implants or metallic devices in the head
* Any history of drug or alcohol abuse
* Presence of cardiac pacemaker
* Generalized CSWS

All study patients will be enrolled for treatment with TMS to see if this modality of treatment has any effect on SWI on CSWS.

Additional exclusions are:

* Adults unable to consent
* Pregnant women
* Prisoners
* Wards of the state
* Non English speaking subjects and families

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Spike-Wave Index (SWI) on EEG during sleep following one time 10 minutes of TRPMS-ECA (epileptogenic cortical area) stimulation | After one single 10 minute stimulation
  The Investigators will assess if treatment had any effect on SWI. SWI is measured on EEG during sleep and is defined as percentage of time during sleep where epileptiform discharges are noted. CSWS is defined as SWI of ≥ 85% during sleep. First 30 minutes of sleep will be scored for comparison of pre and post stimulation.

SECONDARY OUTCOMES:
Duration of sustainability (hours) of change in SWI achieved post stimulation | After one single 10 minute stimulation
  The investigator will assess how long of a change in SWI is achieved post stimulation. This will be monitored on EEG during sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Lalit Bansal, M.D., Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Veggiotti P, Pera MC, Teutonico F, Brazzo D, Balottin U, Tassinari CA. Therapy of encephalopathy with status epilepticus during sleep (ESES/CSWS syndrome): an update. Epileptic Disord. 2012 Mar;14(1):1-11. doi: 10.1684/epd.2012.0482. PMID 22426353
- [Result] Rossini PM, Rossi S. Transcranial magnetic stimulation: diagnostic, therapeutic, and research potential. Neurology. 2007 Feb 13;68(7):484-8. doi: 10.1212/01.wnl.0000250268.13789.b2. PMID 17296913
- [Result] Chen R, Cros D, Curra A, Di Lazzaro V, Lefaucheur JP, Magistris MR, Mills K, Rosler KM, Triggs WJ, Ugawa Y, Ziemann U. The clinical diagnostic utility of transcranial magnetic stimulation: report of an IFCN committee. Clin Neurophysiol. 2008 Mar;119(3):504-532. doi: 10.1016/j.clinph.2007.10.014. Epub 2007 Dec 11. PMID 18063409
- [Result] Chen R, Spencer DC, Weston J, Nolan SJ. Transcranial magnetic stimulation for the treatment of epilepsy. Cochrane Database Syst Rev. 2016 Aug 11;(8):CD011025. doi: 10.1002/14651858.CD011025.pub2. PMID 27513825
- [Result] P41 - 1877 Low-frequency repetitive transcranial magnetic stimulation (r-TMS) treatment in children with refractory focal epilepsy: two case reports Thordstein, M et al. European Journal of Paediatric Neurology 2013, Volume 17 , S65
- See also: Transcranial Brain Stimulation With Rapidly Spinning High-Field Permanent Magnets — https://ieeexplore.ieee.org/document/7473846

DOCUMENTS (1):
  • Informed Consent Form (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/30/NCT04034030/ICF_000.pdf